CLINICAL TRIAL: NCT02825212
Title: Efficacy of All-Oral Anti-Viral Therapy for Symptomatic Hepatitis C Virus Infection-Related Cryoglobulinemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Peter Gorevic, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-2282; IN-US-337-1716 (Other: Gilead Sciences)
Record Dates: First submitted 2016-07-03; First posted 2016-07-07 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis C; Cryoglobulinemia
Keywords: Hepatitis C; Cryoglobulinemia
MeSH Terms: conditions — Hepatitis C; Cryoglobulinemia | interventions — ledipasvir, sofosbuvir drug combination; sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Participant with Symptomatic Hepatitis C Virus Infection-Related Cryoglobulinemia (Experimental): Participants treated with either Harvoni or Epclusa
  * Harvoni 90mg/400 mg FDC once daily. Subjects will take 1 tablet daily with or without food.
  * Epclusa 400mg/100mg 400mg/100mg FDC once daily
  Interventions: Drug: Harvoni; Drug: Epclusa

INTERVENTIONS:
Drug: Harvoni — 12 weeks for naïve subjects or non-cirrhotic treatment experienced subjects; or 24 weeks for treatment experienced subjects with cirrhosis
  Other Names: Ledipasvir/Sofosbuvir; LDV/SOF FDC
Drug: Epclusa — once daily for 12 weeks (naïve subjects, non-cirrhotic treatment experienced or treatment experienced subjects with compensated cirrhosis) for genotype 1-6 subjects.
  Other Names: Sofosbuvir/Velpatasvir

SUMMARY:
10 patients with chronic genotype 1 HCV infection and mixed cryoglobulinemia will be treated with Ledipasvir/Sofosbuvir 90mg/400 mg FDC once daily for 12 weeks (naïve subjects or non-cirrhotic treatment experienced subjects) or 24 weeks (treatment experienced subjects with cirrhosis).

The researchers anticipate that approximately 20% of subjects may have cirrhosis.

DETAILED DESCRIPTION:
The treatment of extrahepatic disease manifestations of HCV has largely paralleled that of hepatic disease. Interferon was reported to have efficacy for MC even before linkage of the syndrome to HCV in 1989, and successful combination therapy with ribavirin was found to eliminate virus and lead to the resolution of immunologic abnormalities associated with extrahepatic disease. In addition, ~75% of HCV-associated indolent asymptomatic lymphoproliferative diseases remit with successful antiviral therapy. However, in many instances, MC (notably cutaneous vasculitis) will relapse with recurrence of virus, and may occasionally persist even after clearance. In particular, side effects of Interferon alpha, including the uncovering of frank autoimmune disease, theoretically may mitigate response of extrahepatic disease to treatment. Peg-interferon increased the response rate of MC, and decreased the duration of treatment, but side effects remained problematic.

An alternative approach to the treatment of MC has been the use of immunomodulatory agents. In particular, B-cell expansion in peripheral blood and in lymphoid follicles in the liver prevalent amongst HCV-infected persons provided a rationale for the use of depletion as a therapeutic strategy. Rituximab (anti-CD20) monotherapy has been used mostly for treatment failures/intolerance or in the setting NHL, and has yielded response rates in the setting of involvement of skin (73%); MPGN (70%); joint (53%); and nerve (36%). However, this monoclonal antibody (MAb) has the potential to form immune-complexes with mixed cryoglobulin RF and cause clinical vasculitis in patients with high cryocrits, and may raise the HCV RNA level in rare patients, causing cytotoxicity. Following Rituximab with Peg-IFN plus ribavirin achieved greater than a 60% complete response (CR) in patients resistant to combination treatment alone. Other approaches include the use of Aldesleukin, an inducer of regulatory T-cell activity, MAbs targeted to specific B-cell subsets or costimulatory signal molecules (e.g. BAFF) or agents inhibiting the interaction of HCV core antigen with C1q in cryoprecipitates via the receptor for the globular domain of C1q (gC1qR).

The development of low molecular weight inhibitors of the non-structural proteins (NSPs) elaborated by HCV, in particular 5A, 5B nucleoside and non-nucleoside polymerase inhibitors, and inhibitors of 3/4A serine proteases; to selectively inhibit HCV replication has raised the prospect of "all-oral" treatment for both hepatic and extrahepatic manifestations of disease. However, the use of first generation direct-acting antiviral agents (Telaprevir® and Boceprevir® linear NS3/4A protease inhibitors) was limited by frequent escape mutants, efficacy restricted to genotype-1, need to retain protocols including PegIFN and ribavirin, potential for significant drug interactions, and serious side effects. In a trial of combination therapy including Telaprevir® for 13 patients with MC, all had significant AEs, including asthenia (92%), anemia (84%), neutropenia and bacterial infection (54%). Approval of an uridine nucleoside analogue that selectively inhibits HCV NS5B RNA-dependent RNA polymerase (Sofosbuvir) by the FDA late 2013 has led to proof-of-concept trials in which combination all-oral therapy has proven effective for both genotype 1 and other genotypes, with a number of other regimens under development. In particular, the combination of Sobosbuvir (SOF) and Ledipasvir (LDV) has been reported to have almost universal efficacy in a 12 week regimen for genotype 1, and the combination of SOF and Ribavirin (RBV) for genotypes 2-6 in a 24 week regimen. However, persistence of cryoglobulinemia even after viral clearance with the newer regimens has also raised the question of whether longer treatment regimens may be appropriate in the setting of significant extrahepatic disease. Thus, the timing is right to initiate a trial of all-oral treatment to rigorously evaluate the effect on extrahepatic disease, and to re-establish the efficacy of antiviral therapy in halting the direct and indirect role of HCV in driving autoimmune disease and lymphoproliferation. Using an interferon-sparing regimen to treat patients with HCV-related cryoglobulinemia will help answer the question as to whether immunomodulating therapy plays a role at all in eradicating cryoglobulins long-term, and whether antiviral therapy alone is adequate. If the latter, appreciable morbidity and mortality may be saved in avoiding treating these potentially sick, often cirrhotic patients, with immunomodulatory therapies.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

1. Willing and able to provide written informed consent
2. Male or female, age ≥18 years
3. HCV RNA ≥ 15 IU/mL at Screening
4. HCV genotype 1
5. Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy
6. Classification as treatment naïve or treatment experienced:

   1. Treatment naïve is defined as having never been exposed to approved or experimental HCV-specific direct-acting antiviral agents or prior treatment of HCV with interferon or ribavirin or DAAs (except for SOF-containing regimens).
   2. Treatment experienced is defined as prior treatment failure or relapse to a regimen containing interferon either with or without RBV or DAAs (except for SOF-containing regimens) that was completed at least 8 weeks prior to Baseline/Day 1.

   The subject's medical records must include sufficient detail of prior virologic failure to allow for categorization of prior response, as either:
   1. Non-Responder: Subject did not achieve undetectable HCV RNA levels while on treatment, or
   2. Relapse/Breakthrough: Subject achieved undetectable HCV RNA levels during treatment or within 4 weeks of the end of treatment but did not achieve SVR.
7. Cirrhosis determination (approximately 20% of subjects may have cirrhosis) a. Cirrhosis is defined as any one of the following:

   i) Any previous liver biopsy showing cirrhosis (e.g., Metavir score = 4 or Ishak score ≥5) ii) FibroMeter® score >0.442 or an AST:platelet ratio index (APRI) >2 during Screening iii) Fibroscan with a result of >12.5 kPa at any time prior to or during screening.

   b. Absence of cirrhosis is defined as any one of the following: i) Liver biopsy within 2 years of Screening showing absence of cirrhosis ii) FibroMeter® score <0.442 or APRI ≤ 1 performed during Screening iii) Fibroscan with a result of ≤12.5 kPa within 6 months of Baseline/Day 1 Fibroscan results will supersede FibroMeter® /APRI; liver biopsy results will supersede Fibrotest® /APRI or Fibroscan results and be considered definitive.
8. Liver imaging (ultrasound, CT scan or MRI) within 6 months of screening is required in patients with cirrhosis to exclude hepatocellular carcinoma (HCC)
9. Presence of MC vasculitis (please see criteria on the note below).
10. Null or partial response to previous therapies for MC, including corticosteroids, cytotoxic agents (cyclophosphamide, azathioprine), hydroxychloroquine, methotrexate, mono- or combination therapy with IFNα/PEG-IFN and ribavirin, and/or CD20 depletion with Rituximab. a. Patients can be on ongoing treatment with one of the drugs described above at inclusion unless there is significant DDI.
11. Subjects has the following laboratory parameters at screening:

    1. ALT <10 x the upper limit of normal (ULN)
    2. AST <10 x ULN
    3. Adequate bone marrow function as indicated hematologic parameters listed below and/or bone marrow cellularity >60-70% average for age.

    i. WBC >1500 /uL ii.Platelets > 50,000/uL

    d) Direct bilirubin >2 x ULN e) INR >1.5 x ULN unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
12. Females of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Baseline/Day 1 prior to treatment.
13. Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception.
14. Lactating females must agree to discontinue nursing before the study drug is administered.
15. Subject must be of generally good health, with the exception of chronic HCV infection, as determined by the Investigator.
16. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Note: Definition of Mixed Cryoglobulinemia (patients must meet one of the five overlapping syndromes listed below and the presence of cold-precipitable immune complexes in blood on two different occasions.

* Clinical evidence of cryoglobulinemia, overlapping syndromes:

  1. Cutaneous vasculitis (Raynaud's phenomenon, purpura, skin ulcers, livedo, acrocyanosis)
  2. Glomerulonephritis (hypertension, hematuria, nephrotic syndrome)
  3. Arthropathy (arthralgias, arthritis)
  4. Neuropathy (peripheral and/or central nervous system, distal sensorimotor, mononeuritis multiplex)
  5. Sicca syndrome (xerostomia, xerophthalmia)

     Other factors that will be assessed / recorded in patients with MC will be:

  1. Associated laboratory abnormalities including:
* Positive HCV serology (recombinant immunoblot assay), viral nucleic acid quantitation diagnostic for HCV infection, and reflex genotyping.
* Evidence of glomerulonephritis, including an active urinary sediment, hypoalbuminemia (albumin <3gm/dL) and/or significant proteinuria (>300mg/day).
* Abnormal nerve conduction testing. 2. Pathologic evidence of cryoglobulinemia including:
* Leukocytoclastic vasculitis.
* Membranoproliferative glomerulonephritis.
* Vasculopathy and/or mononuclear cell infiltrates on sural nerve biopsy.
* Lip biopsy suggestive for Sjogren's syndrome. 3. Laboratory evidence of cryoglobulinemia including:
* Characterization of cryoprecipitable material in serum by immunofixation, cryocrit, and/or quantitation of protein.
* Associated immunological abnormalities, such as depressed levels of complement, elevated titers of rheumatoid factor, abnormal immunoglobulin quantitations, and serum immunofixation carried out on serum and/or isolated cryoglobulins.

  4. Laboratory evidence of B-cell clonality, including:
* IgMk determined by immunofixation of serum and/or cryoglobulin, and kappa excess >2.65:1 on Free Light Chain (FLC) assay

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gorevic, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dammacco F, Sansonno D. Therapy for hepatitis C virus-related cryoglobulinemic vasculitis. N Engl J Med. 2013 Sep 12;369(11):1035-45. doi: 10.1056/NEJMra1208642. No abstract available. PMID 24024840
- [Background] Damoiseaux J. The diagnosis and classification of the cryoglobulinemic syndrome. Autoimmun Rev. 2014 Apr-May;13(4-5):359-62. doi: 10.1016/j.autrev.2014.01.027. Epub 2014 Jan 11. PMID 24424176
- [Background] Jacobson IM, Cacoub P, Dal Maso L, Harrison SA, Younossi ZM. Manifestations of chronic hepatitis C virus infection beyond the liver. Clin Gastroenterol Hepatol. 2010 Dec;8(12):1017-29. doi: 10.1016/j.cgh.2010.08.026. Epub 2010 Sep 24. PMID 20870037
- [Background] Giordano TP, Henderson L, Landgren O, Chiao EY, Kramer JR, El-Serag H, Engels EA. Risk of non-Hodgkin lymphoma and lymphoproliferative precursor diseases in US veterans with hepatitis C virus. JAMA. 2007 May 9;297(18):2010-7. doi: 10.1001/jama.297.18.2010. PMID 17488966
- [Background] Ko HM, Hernandez-Prera JC, Zhu H, Dikman SH, Sidhu HK, Ward SC, Thung SN. Morphologic features of extrahepatic manifestations of hepatitis C virus infection. Clin Dev Immunol. 2012;2012:740138. doi: 10.1155/2012/740138. Epub 2012 Aug 5. PMID 22919404
- [Background] Dispenzieri A, Gorevic PD. Cryoglobulinemia. Hematol Oncol Clin North Am. 1999 Dec;13(6):1315-49. doi: 10.1016/s0889-8588(05)70129-5. PMID 10626153
- [Background] Gorevic PD. Rheumatoid factor, complement, and mixed cryoglobulinemia. Clin Dev Immunol. 2012;2012:439018. doi: 10.1155/2012/439018. Epub 2012 Aug 26. PMID 22956968
- [Background] Wilson LE, Widman D, Dikman SH, Gorevic PD. Autoimmune disease complicating antiviral therapy for hepatitis C virus infection. Semin Arthritis Rheum. 2002 Dec;32(3):163-73. doi: 10.1053/sarh.2002.37277. PMID 12528081
- [Background] Saadoun D, Resche Rigon M, Thibault V, Longuet M, Pol S, Blanc F, Pialoux G, Karras A, Bazin-Karra D, Cazorla C, Vittecoq D, Musset L, Decaux O, Ziza JM, Lambotte O, Cacoub P. Peg-IFNalpha/ribavirin/protease inhibitor combination in hepatitis C virus associated mixed cryoglobulinemia vasculitis: results at week 24. Ann Rheum Dis. 2014 May;73(5):831-7. doi: 10.1136/annrheumdis-2012-202770. Epub 2013 Apr 20. PMID 23606708
- [Background] Kowdley KV, Gordon SC, Reddy KR, Rossaro L, Bernstein DE, Lawitz E, Shiffman ML, Schiff E, Ghalib R, Ryan M, Rustgi V, Chojkier M, Herring R, Di Bisceglie AM, Pockros PJ, Subramanian GM, An D, Svarovskaia E, Hyland RH, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Pound D, Fried MW; ION-3 Investigators. Ledipasvir and sofosbuvir for 8 or 12 weeks for chronic HCV without cirrhosis. N Engl J Med. 2014 May 15;370(20):1879-88. doi: 10.1056/NEJMoa1402355. Epub 2014 Apr 10. PMID 24720702
- [Background] Afdhal N, Zeuzem S, Kwo P, Chojkier M, Gitlin N, Puoti M, Romero-Gomez M, Zarski JP, Agarwal K, Buggisch P, Foster GR, Brau N, Buti M, Jacobson IM, Subramanian GM, Ding X, Mo H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Mangia A, Marcellin P; ION-1 Investigators. Ledipasvir and sofosbuvir for untreated HCV genotype 1 infection. N Engl J Med. 2014 May 15;370(20):1889-98. doi: 10.1056/NEJMoa1402454. Epub 2014 Apr 11. PMID 24725239
- [Background] Levo Y, Gorevic PD, Kassab HJ, Tobias H, Franklin EC. Liver involvement in the syndrome of mixed cryoglobulinemia. Ann Intern Med. 1977 Sep;87(3):287-92. doi: 10.7326/0003-4819-87-3-287. PMID 900672
- [Background] Diagnosis and treatment of HCV-related mixed cryoglobulinemia over the last decade at a Liver Referral Center Ando, Y, Gorevic, PD, Schiano TD. Hepatology 58 2013 : 1443 abstract
- [Background] Naarendorp M, Kallemuchikkal U, Nuovo GJ, Gorevic PD. Longterm efficacy of interferon-alpha for extrahepatic disease associated with hepatitis C virus infection. J Rheumatol. 2001 Nov;28(11):2466-73. PMID 11708420
- [Background] Levine JW, Gota C, Fessler BJ, Calabrese LH, Cooper SM. Persistent cryoglobulinemic vasculitis following successful treatment of hepatitis C virus. J Rheumatol. 2005 Jun;32(6):1164-7. PMID 15940780
- [Background] Chen AY, Zeremski M, Chauhan R, Jacobson IM, Talal AH, Michalak TI. Persistence of hepatitis C virus during and after otherwise clinically successful treatment of chronic hepatitis C with standard pegylated interferon alpha-2b and ribavirin therapy. PLoS One. 2013 Nov 21;8(11):e80078. doi: 10.1371/journal.pone.0080078. eCollection 2013. PMID 24278242
- [Background] Piluso A, Giannini C, Fognani E, Gragnani L, Caini P, Monti M, Petrarca A, Ranieri J, Urraro T, Triboli E, Laffi G, Zignego AL. Value of IL28B genotyping in patients with HCV-related mixed cryoglobulinemia: results of a large, prospective study. J Viral Hepat. 2013 Apr;20(4):e107-14. doi: 10.1111/jvh.12017. Epub 2012 Dec 4. PMID 23490377
- [Background] Russi S, Sansonno D, Mariggio MA, Vinella A, Pavone F, Lauletta G, Sansonno S, Dammacco F. Assessment of total hepatitis C virus (HCV) core protein in HCV-related mixed cryoglobulinemia. Arthritis Res Ther. 2014 Mar 18;16(2):R73. doi: 10.1186/ar4513. PMID 24636026
- [Background] Sansonno D, Tucci FA, Ghebrehiwet B, Lauletta G, Peerschke EI, Conteduca V, Russi S, Gatti P, Sansonno L, Dammacco F. Role of the receptor for the globular domain of C1q protein in the pathogenesis of hepatitis C virus-related cryoglobulin vascular damage. J Immunol. 2009 Nov 1;183(9):6013-20. doi: 10.4049/jimmunol.0902038. Epub 2009 Oct 14. PMID 19828637
- [Background] Quartuccio L, Isola M, Corazza L, Ramos-Casals M, Retamozo S, Ragab GM, Zoheir MN, El-Menyawi MA, Salem MN, Sansonno D, Ferraccioli G, Gremese E, Tzioufas A, Voulgarelis M, Vassilopoulos D, Scarpato S, Pipitone N, Salvarani C, Guillevin L, Terrier B, Cacoub P, Filippini D, Saccardo F, Gabrielli A, Fraticelli P, Sebastiani M, Tomsic M, Tavoni A, Mazzaro C, Pioltelli P, Nishimoto N, Scaini P, Zignego AL, Ferri C, Monti G, Pietrogrande M, Bombardieri S, Galli M, De Vita S. Validation of the classification criteria for cryoglobulinaemic vasculitis. Rheumatology (Oxford). 2014 Dec;53(12):2209-13. doi: 10.1093/rheumatology/keu271. Epub 2014 Jul 3. PMID 24994905
- [Background] Felson DT, Anderson JJ, Boers M, Bombardier C, Furst D, Goldsmith C, Katz LM, Lightfoot R Jr, Paulus H, Strand V, et al. American College of Rheumatology. Preliminary definition of improvement in rheumatoid arthritis. Arthritis Rheum. 1995 Jun;38(6):727-35. doi: 10.1002/art.1780380602. PMID 7779114
- [Background] Stone JH, Hoffman GS, Merkel PA, Min YI, Uhlfelder ML, Hellmann DB, Specks U, Allen NB, Davis JC, Spiera RF, Calabrese LH, Wigley FM, Maiden N, Valente RM, Niles JL, Fye KH, McCune JW, St Clair EW, Luqmani RA; International Network for the Study of the Systemic Vasculitides (INSSYS). A disease-specific activity index for Wegener's granulomatosis: modification of the Birmingham Vasculitis Activity Score. International Network for the Study of the Systemic Vasculitides (INSSYS). Arthritis Rheum. 2001 Apr;44(4):912-20. doi: 10.1002/1529-0131(200104)44:43.0.CO;2-5. PMID 11318006
- [Background] Ozkok A, Yildiz A. Hepatitis C virus associated glomerulopathies. World J Gastroenterol. 2014 Jun 28;20(24):7544-54. doi: 10.3748/wjg.v20.i24.7544. PMID 24976695
- [Background] Benstead TJ, Chalk CH, Parks NE. Treatment for cryoglobulinemic and non-cryoglobulinemic peripheral neuropathy associated with hepatitis C virus infection. Cochrane Database Syst Rev. 2014 Dec 20;2014(12):CD010404. doi: 10.1002/14651858.CD010404.pub2. PMID 25525951
- [Background] Gragnani L, Fognani E, Piluso A, Boldrini B, Urraro T, Fabbrizzi A, Stasi C, Ranieri J, Monti M, Arena U, Iannacone C, Laffi G, Zignego AL; MaSVE Study Group. Long-term effect of HCV eradication in patients with mixed cryoglobulinemia: a prospective, controlled, open-label, cohort study. Hepatology. 2015 Apr;61(4):1145-53. doi: 10.1002/hep.27623. Epub 2015 Feb 10. PMID 25431357
- [Background] Foulks GN, Forstot SL, Donshik PC, Forstot JZ, Goldstein MH, Lemp MA, Nelson JD, Nichols KK, Pflugfelder SC, Tanzer JM, Asbell P, Hammitt K, Jacobs DS. Clinical guidelines for management of dry eye associated with Sjogren disease. Ocul Surf. 2015 Apr;13(2):118-32. doi: 10.1016/j.jtos.2014.12.001. Epub 2015 Jan 15. PMID 25881996
- [Background] Delli K, Spijkervet FK, Kroese FG, Bootsma H, Vissink A. Xerostomia. Monogr Oral Sci. 2014;24:109-25. doi: 10.1159/000358792. Epub 2014 May 23. PMID 24862599
- [Background] Aletaha D, Landewe R, Karonitsch T, Bathon J, Boers M, Bombardier C, Bombardieri S, Choi H, Combe B, Dougados M, Emery P, Gomez-Reino J, Keystone E, Koch G, Kvien TK, Martin-Mola E, Matucci-Cerinic M, Michaud K, O'Dell J, Paulus H, Pincus T, Richards P, Simon L, Siegel J, Smolen JS, Sokka T, Strand V, Tugwell P, van der Heijde D, van Riel P, Vlad S, van Vollenhoven R, Ward M, Weinblatt M, Wells G, White B, Wolfe F, Zhang B, Zink A, Felson D; EULAR; ACR. Reporting disease activity in clinical trials of patients with rheumatoid arthritis: EULAR/ACR collaborative recommendations. Arthritis Rheum. 2008 Oct 15;59(10):1371-7. doi: 10.1002/art.24123. PMID 18821648
- [Background] Gorevic, PD; "Mixed Cryoglobulinemia Cross-reactive Idiotypes: Structural and Clinical Significance" Cryoglobulinemia & Hepatitis C Infection, Dammacco, F (Editor); Springer Verlag, 2012, p. 99-107.
- [Background] Gorevic PD and Galanakis DK;

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were self referred after discussion with their physicians, enrolled sequentially over a two year period (2016-2018)
Pre-assignment Details: Long recruitment, with part of the problem of finding patients not already on antivirals. The original protocol was for Harvoni, which had been specifically licensed for Hepatitis C Virus genotype 1. Protocol was modified after discussion with Gilead with the licensing of Epclusa, which is active for other genotypes, specifically to be able to include two patients with genotype 2 thus enabling the study to reach full enrollment. Study objective is not to compare medications.
Groups:
- Pts With Hep C Virus Infection-Related Cryoglobulinemia: Participants with Symptomatic Hepatitis C Virus Infection-Related Cryoglobulinemia who were treated with antivirals.
  Antivirals were either Harvoni or Epclusa. Ledipasvir/Sofosbuvir (Harvoni) 90mg/400 mg FDC once daily for 12 weeks (naïve subjects, non-cirrhotic treatment experienced subjects) or 24 weeks (treatment experienced subjects with compensated cirrhosis) for genotype 1 .
  Sofosbuvir/Velpatasvir (Epclusa) 400mg/100mg 400mg/100mg FDC once daily for 12 weeks (naïve subjects, non-cirrhotic treatment experienced or treatment experienced subjects with compensated cirrhosis) for genotype 1-6 subjects.
Period: Overall Study
Arm/Group | Pts With Hep C Virus Infection-Related Cryoglobulinemia
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pts With Hep C Virus Infection-Related Cryoglobulinemia
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 3
  Hispanic | 1
  Asian | 1
  Unknown | 5
Years Since HCV Diagnosis [Mean (Standard Deviation); unit: years] | 16.1 (12.29)
Treatment Naive [Count of Participants; unit: Participants] | 3
Cirrhosis [Count of Participants; unit: Participants] — diagnosed by imaging or biopsy
  Participants | 2
AST levels [Mean (Standard Deviation); unit: U/L] — normal is <40 U/L
  U/L | 74.7 (99.41)
Platelets level [Mean (Standard Deviation); unit: K/uL] — normal 150-450K/uL
  K/uL | 192.7 (73.96)
HCV genotype [Count of Participants; unit: Participants]
  1a | 3
  1b | 5
  2 | 1
  2a | 1
Bilirubin [Mean (Standard Deviation); unit: mg/dL] — normal <1.2 mg/dL
  mg/dL | 0.93 (1.66)
Viral Count [Mean (Standard Deviation); unit: IU/ml] | 78.98 (136.72)
Hepa Score for Fibrosis [Count of Participants; unit: Participants] — Quantitative results of 6 biochemical tests analyzed using a computational algorithm to provide a quantitative surrogate marker (0.0-1.0) for liver fibrosis (METAVIR F0-F4).
  Fibrosis scoring
  <0.21 = Stage F0 - No fibrosis
  0.21 - 0.27 = Stage F0 - F1
  0.27 - 0.31 = Stage F1 - Portal fibrosis
  0.31 - 0.48 = Stage F1 - F2
  0.48 - 0.58 = Stage F2 - Bridging fibrosis with few septa
  0.58 - 0.72 = Stage F3 - Bridging fibrosis with many septa
  0.72 - 0.74 = Stage F3 - F4
  >0.74 = Stage F4 - Cirrhosis
  Participants
    F0-F1 | 2
    F1 | 1
    F1-F2 | 1
    F2 | 1
    F2-F4 | 1
    F3 | 3
    F4 | 1

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virologic Response (SVR)
Description: Number of participants who attain SVR, ie, cleared HCV
Time Frame: 2-4 weeks and 24 weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pts With Hep C Virus Infection-Related Cryoglobulinemia
Number analyzed (Participants) | 10
Participants
  2-4 weeks after treatment | 10
  24 weeks after treatment | 10

2. Primary Outcome: Response in Patients With Mixed Cryoglobulinemia (MC)
Description: Response to medication in patients with MC categorized as either complete response (100% response) vs partial response (50% response).
Time Frame: up to 24 weeks after treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pts With Hep C Virus Infection-Related Cryoglobulinemia
Number analyzed (Participants) | 10
Participants
  Partial Response | 9
  Complete Response | 0
  No Response | 1

ADVERSE EVENTS:
Time Frame: up to 24 weeks after treatment
Arm/Group | Pts With Hep C Virus Infection-Related Cryoglobulinemia
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pts With Hep C Virus Infection-Related Cryoglobulinemia (N=10)
Herpes Zoster (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pts With Hep C Virus Infection-Related Cryoglobulinemia (N=10)
Increased fatigue (General disorders) | 4
nausea and abdominal pain (Gastrointestinal disorders) | 3
Urinary frequency and/or dysuria (Renal and urinary disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT02825212/Prot_SAP_000.pdf